CLINICAL TRIAL: NCT03006003
Title: The Assessment of Osteoporosis Treatment in Post-menopausal Women
Brief Title: Osteoporosis Treatment in Post-menopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE16256A
Record Dates: First submitted 2016-12-16; First posted 2016-12-30 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2018-01

CONDITIONS: Depressive Syndrome
Keywords: Osteoporosis; Raloxifene; Central nervous disorders
MeSH Terms: conditions — Depressive Disorder; Osteoporosis | interventions — Raloxifene Hydrochloride; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Raloxifene group (Experimental): Raloxifene treatment
  Interventions: Drug: Raloxifene
- Comparator group (Active Comparator): Alendronate treatment
  Interventions: Drug: Alendronate
- Control group (No Intervention): To refuse anti-osteoporosis treatment

INTERVENTIONS:
Drug: Raloxifene — Raloxifene tratment more than 4 weeks
  Other Names: Evista
  Arms: Raloxifene group
Drug: Alendronate — Alendronic acid 70mg with Colecalciferol 70mcg
  Other Names: FOSAMAX PLUS
  Arms: Comparator group

SUMMARY:
The study will be conducted to assess the depressive symptoms and related markers in the postmenopausal female after anti-osteoporosis treatment.

DETAILED DESCRIPTION:
Fracture is one of the important complications in female. Osteoporosis should be treated in postmenopausal female due to high risk of fracture. Recently, there have been many classes of medications developed for preventing bone loss. Raloxifene, an oral form of anti-osteoporosis medication, has been reported to improved central nervous disorders. Therefore, this study is designed to assess the depressive symptoms and related markers in the postmenopausal female after anti-osteoporosis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female
* Osteoporosis

Exclusion Criteria:

* Psychological disorders

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Brain-derived neurotrophic factor | 3 months
  Serum brain-derived neurotrophic factor (BDNF) Levels

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor | 1 year
  Serum brain-derived neurotrophic factor (BDNF) Levels
Vascular cell adhesion molecule-1 | 3 months
  Serum vascular cell adhesion molecule-1 (VCAM-1) levels
Orexin-A | 3 months
  Serum Orexin-A levels
Body components | 3 months
  Fat tissue ratio
Zung self-rating depression scale | 3 months
  Questionnaire for depressive symptoms
5-Item Geriatric Depression Scale | 3 months
  Questionnaire for Cognitive assessment
The Mini Mental State Examination (MMSE) | 3 months
  Questionnaire for Cognitive assessment
The Barthel index | 3 months
  Questionnaire for Cognitive assessment
Instrumental Activities of Daily Living (IADL) | 3 months
  Questionnaire for Cognitive assessment
ankle-brachial index | 3 months
  Peripheral artery disease assessment

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - outpatient clinic of the Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No